CLINICAL TRIAL: NCT02987127
Title: Prospective Study of Frontline Helicobacter Pylori Eradication Therapy in the Treatment of Early-stage Extragastric Mucosa-associated Lymphoid Tissue Lymphoma
Brief Title: Prospective Study of Frontline H Pylori Eradication in the Treatment of Early-stage Extragastric MALT Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511025MINC
Record Dates: First submitted 2016-12-01; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Mucosa-Associated Lymphoid Tissue Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Gastric low-grade mucosa-associated lymphoid tissue lymphoma (MALToma) is associated with Helicobacter pylori (HP) infection, and around 70% of these tumors can be cured by HP eradication therapy (HPE). However, the role of antibiotics in the frontline treatment of extragastric MALToma remains unclear. In addition to anecdotal case reports showing histologic regression of extragastric MALTomas after antibiotics, our explorative study found that frontline HPE (clarithromycin, amoxicillin, and omeprazole) resulted in complete remission (CR) in this subgroup patients (2 salivary gland, 1 lung, 1 colon, and 4 ocular adnexal MALToma [OAML]). Interestingly, two patients with OAML who do not respond to Chlamydia psittaci (CP) eradication using doxycycline achieved CR after HPE. These findings suggest that bacterial infections, including HP, may be involved in the lymphomagenesis of these extragastric MALTomas. Our preliminary results also revealed that 5 (23.8%) of 21 HP-negative gastric MALToma patients achieved CR after HPE, indicating that antibiotics may also have ability to eradicate non-HP bacteria. Based on our preliminary findings and the indolent biologic behavior of MALToma, it is reasonable to use frontline HPE in the treatment of early-stage low-grade extragastric MALToma.

DETAILED DESCRIPTION:
Through a prospective trial of frontline HPE in the treatment of early-stage extragastric MALToma, investigators will evaluate and investigate the following issues:

1. The CR and partial remission (PR) rate for antibiotics as 1st-line therapy for stage IE and stage IIE extragastric MALToma
2. The durability of CR and PR (relapse-free survival) after antibiotics treatment (HPE) in early-stage extragastric MALToma
3. The assessment of the evidence of bacterial infection, such as HP, in extragastric MALToma.
4. The identification of potential biomarkers that help us predict whether extragastric MALToma can respond to frontline HPE.

ELIGIBILITY:
Inclusion Criteria:

1. The patients must have histologically confirmed low-grade mucosa-associated
2. lymphoid tissue lymphoma of extragastric sites.
3. Patients must have evaluable disease by physical examination, endoscopy (also include colonfibroscopy, and bronchoscopy) or computed tomography.
4. Patients must receive examination of documented HP infection or not before treatment, which will be evaluated by the following tests: histology, rapid urease test (CLO-test), C-13 urease breath test and serology.
5. Patients must have either stage IE or IIE-1 disease, according to an adaptation of the Ann Arbor staging system modified by Musshoff for primary extranodal lymphoma.
6. Patients must have signed the informed consent and agree to provide achieved pathologic material for immunohistochemical staining of BCL10, NF-KB, BAFF, CagA, CagA-signaling molecules, for fluorescence in situ hybridization study for t(11;18)(q21;q21)/API2-MALT1 and t(14;18)(q32;q21)/IGH-MALT1 determination, and for PCR of Chlamydia psittaci and Borrelia burgdorferi.
7. Patients must have signed the informed consent and agree to provide achieve blood samples for CYP2C19 genetic polymorphisms evaluation and potential serum molecular studies, such as serum BAFF level

Exclusion Criteria:

1. In the diagnosis of the disease over the past five years with a history of other cancers but non-melanoma skin cancer, breast and cervical carcinoma in situ carcinoma in situ (leafy or tubular) can still meet the conditions of admission to this case study
2. Patients receiving chemotherapy or radiotherapy of nodules outside the low-grade malignant lymphoma, but has not yet been cured, the excluded
3. The second more, and not in the lymph nodes adjacent to the tumor (IIE-2 period or more), the excluded
4. The state can not afford this clinical cardiopulmonary ㄧ inspection after the test series, the excluded
5. suffering from primary gastric outside MALToma before and had received chemotherapy or radiation therapy in patients of.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Extragastric mucosa-associated lymphoid tissue lymphoma
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The complete and partial remission rate for antibiotics as 1st-line therapy for stage IE-IIE1 extragastric MALT lymphoma. | 5 years
  The complete remission rate and partial remission rate for antibiotics (HP eradicaiton) as 1st-line therapy for early-stage extragastric MALT lymphoma

SECONDARY OUTCOMES:
The overall survival of early-stage extragastric MALT lymphoma patients who received frontline HP eradication therapy | 5 years
The assessment of the evidence of bacterial infection in all extragstric MALT lymphoma | 5 years
The usefulness of pattern of NF-κB, BCL10, BAFF, API2-MALT1, and IgH-MALT1 by IHC staining or FISH in prospectively predicting the antibiotics responsiveness of extragastric MALT lymphoma | 5 years
The relapse-free survival of early-stage extragastric MALT lymphoma patients who received antibiotics as 1st-line therapy | 5 years

OTHER OUTCOMES:
The complete remission rate and durability of second-line chemotherapy with chlorambucil plus prednisolone for progressive disease after frontline HP eradication therapy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hsin Kuo, M.D.,Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No